CLINICAL TRIAL: NCT05929196
Title: Feasibility Evaluation - Blood Glucose Level Monitoring by Microwave Metamaterial Sensor in Blood Samples.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Czech Technical University in Prague (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: FBMI_MTM_sensor; 1/2023/LOK (Other: Oblastní nemocnice Kladno)
Record Dates: First submitted 2023-05-05; First posted 2023-07-03 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Diabetes
Keywords: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Blood sample donator (Experimental): The participant donates approximately 5 ml of blood sample.
  Interventions: Diagnostic Test: In vitro full blood diagnostic test.

INTERVENTIONS:
Diagnostic Test: In vitro full blood diagnostic test. — Participant will donate approximately 5 ml blood sample. Later in a laboratory the sample will be processed in the microwave metamaterial sensor for non invasive blood glucose monitoring and standard biochemical analyzer. Specific dielectric properties and scattering parameters will be measured for blood glucose level determination.

SUMMARY:
The goal of this clinical trial is to test microwave metamaterial glucose sensor on blood samples. It means to compare the results of glucose values obtained by microwave metamaterial sensor and by standard biochemical analyzer.

DETAILED DESCRIPTION:
Participants will include physiological and pathological populations. Participants donate approximately 5 ml of blood sample. Three sample tubes will be collected from ten adult participants. In the first test tube, the blood glucose content will be determined by a validated biochemical analyzer (Roche, Switzerland). In the remaining volume of the blood sample, the dielectric parameters (relative permittivity and conductivity) will be estimated using a coaxial probe (Keysight, USA). Microwave metamaterial sensors with 5, 7 and 9 unit cells will be loaded with blood samples and the specific scattering matrices will be obtained using a vector network analyzer. The main monitored outcome measure will be the phase of parameter S21.

ELIGIBILITY:
Inclusion Criteria:

* blood glucose can be measured with standard biochemical analyzer

Exclusion Criteria:

* minimum age limit 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2023-07-12 (Actual); Primary Completion 2023-07-17 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Phase shift of scattering parameter S21 | When blood sample is filled into sensor chamber within 24 hours from blood collection.
  The proposed microwave sensor uses a section of planar metamaterial transmission line operating at GHz frequencies. The speed of electromagnetic wave propagation through the sample is affected by the concentration of glucose. The delay can be expressed in degrees (°) as the phase of the complex S21 parameter.
Blood glucose concentration | When blood sample is processed in biochemical analyzer within 24 hours from blood collection.
  Molar mass of glucose dissolved in liquid blood sample expressed as molar concentration (mmol/l).
Blood sample specific electrical conductivity | When blood sample is presented into the co-axial probe container within 24 hours from blood collection.
  The specific electrical conductivity (S/m) of the blood samples will be measured using a coaxial probe.
Blood sample relative permittivity | When blood sample is presented into the co-axial probe container within 24 hours from blood collection.
  The relative permittivity (-) of the blood samples will be measured using a coaxial probe.

SECONDARY OUTCOMES:
Sensor sensitivity | After primary data acqiusition.
  Present the relation between the value of he Phase shift of scattering parameter S21 and Blood glucose concentration.
Mathematical model of blood glucose dependence on blood dielectric parameters | After primary data acqiusition.
  The mathematical model describing which combination of dielectric parameter values (specific electrical conductivity and relative permittivity) corresponds to the certain blood glucose level.

CONTACTS AND LOCATIONS:
Overall Officials: Luděk Šprongl, Ing., Principal Investigator — Regional hospital in Kladno; Lukáš Malena, Ing., Principal Investigator — Czech Technical University in Prague; David Vrba, doc., Principal Investigator — Czech Technical University in Prague
Locations (1):
- Oblastní nemocnice Kladno, a.s., Kladno, Central Bohemia, Czechia